CLINICAL TRIAL: NCT05922722
Title: Clarifying Misbeliefs About Hydroxychloroquine (HCQ): Developing an Individualized Decision Aid for Diverse Patients With Lupus (HCQ-IDEAL)
Brief Title: Clarifying Misbeliefs About Hydroxychloroquine: Developing a Decision Aid for Patients With Lupus
Acronym: HCQ-IDEAL
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0846; Protocol Version 5/23/23 (Other: UW Madison); SMPH/MEDICINE/RHEUMATOL (Other: UW Madison)
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Lupus
Keywords: hydroxychloroquine
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with lupus
  Interventions: Other: Decision-making tool; Other: Questionnaire

INTERVENTIONS:
Other: Decision-making tool — The shared decision-making tool is a paper tool or an electronic version which will be available in the clinics for clinic team's use.
Other: Questionnaire — Questionnaire to assess participant's understanding of the decision-making tool

SUMMARY:
The purpose of this research study is to collect information from lupus patients about their experience with a tool that informs patients about the benefits vs. harms of a medication such as hydroxychloroquine. The main question it aims to answer is whether the decision-making tool will increase medication adherence.

Participants will be asked to complete questionnaires that assess their understanding of the decision-making tool.

DETAILED DESCRIPTION:
This study will be no different from a routine lupus or lupus nephritis clinic visit. During the same visit that a participant routinely does for lupus with their healthcare team, a healthcare team member will discuss the tool that elaborates the benefits vs. risks of lupus medications such as hydroxychloroquine. Participants will complete questionnaires that assesses their understanding of the medication (hydroxychloroquine) before and after they complete the discussion regarding the medication using the tool with the healthcare team member.

Study team members will study the data collected to answer research questions. They will analyze the data and plan better steps improve care quality in lupus.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* validated SLE diagnosis
* no absolute contraindication to HCQ (e.g., retinopathy)
* prior HCQ therapy for at least 3-6 months

Exclusion Criteria:

* participants with other autoimmune diseases
* participants who are not taking HCQ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with validated lupus diagnosis on Hydroxychloroquine (HCQ)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence | Baseline to 3 months
  Compare mean adherence at baseline and three months after completing the intervention. Mean adherence will be measured using the proportion of days covered (PDC). PDC is calculated using prescription refill data (PDC = Sum of days covered/number of days in the observation period)
Change in medication adherence - participant reported | Baseline to 3 months
  Compare mean adherence at baseline and three months after completing the intervention. Mean adherence will be measured using participant self-report (adherence = 80% prescriptions refilled)
Change in medication adherence - blood levels | Baseline to 3 months
  Compare mean adherence at baseline and three months after completing the intervention. Mean adherence will be measured using blood levels (adherence = 500 ng/ml or higher)
Change in proportion of adherent participants | Baseline to 6 months
  Compare the proportion of adherent patients (Adherence = PDC ≥ 80%) at baseline v 6 months after completing intervention
Change in proportion of adherent participants - participant reported | Baseline to 6 months
  Compare the proportion of adherent patients (Adherence = 80% prescription refills) at baseline v 6 months after completing intervention
Change in proportion of adherent participants - blood levels | Baseline to 6 months
  Compare the proportion of adherent patients through blood levels (Adherence = 500 ng/ml or higher) at baseline v 6 months after completing intervention

SECONDARY OUTCOMES:
Change in decisional conflict scores | Baseline to 6 months
  Decisional conflict scores range from 0 (best) to 1 (worst) with 0.25 as an indicator of residual decisional conflict.
Assess participant satisfaction with decision-making tool | Post-intervention, on average 6 months
  Participant satisfaction using a Likert scale 0-7 (7=most satisfied)
Intervention completion | Duration of study, up to 12 months
  Total number of visits with participants completing the intervention during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Shivani Garg, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No